CLINICAL TRIAL: NCT03661385
Title: A Randomised Controlled Trial of Nitric Oxide Administration During Cardiopulmonary Bypass in Infants Undergoing Arterial Switch Operation for Repair of Transposition of the Great Arteries
Brief Title: Nitric Oxide During Bypass for Arterial Switch Operation
Acronym: NASO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Murdoch Childrens Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 38017; ACTRN12618000089235p (Registry Identifier: ANZCTR)
Record Dates: First submitted 2018-09-04; First posted 2018-09-07 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Low Cardiac Output Syndrome; Transposition of Great Vessels
Keywords: Cardiopulmonary bypass; Congenital heart disease; Low cardiac output syndrome; Nitric oxide; Transposition of Great Arteries; Arterial switch operation
MeSH Terms: conditions — Cardiac Output, Low; Transposition of Great Vessels; Heart Defects, Congenital | interventions — Nitric Oxide

STUDY DESIGN:
Intervention Model Description: Double blinded, randomised controlled, parallel study comparing an intervention with a control.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Perfusionist (operating bypass) is unblinded to randomisation. They will randomize patient in a computer base (REDcap).Randomization is blinded to all other staff and the nitric oxide container is draped. Nitric oxide container will be attached in all cases.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intervention arm (Active Comparator): • Intervention arm will receive nitric oxide 20 parts per million (ppm) into the oxygenator of a cardio-pulmonary bypass circuit
  Interventions: Drug: Nitric Oxide
- Control arm (No Intervention): Control arm will not receive nitric oxide, they will receive standard bypass as per local policy

INTERVENTIONS:
Drug: Nitric Oxide — Addition of nitric oxide 20ppm into bypass circuit
  Arms: Intervention arm

SUMMARY:
This trial will test if adding nitric oxide (NO) gas to the cardiopulmonary bypass (CPB) circuit in infants undergoing an arterial switch operation (ASO) for Transposition of the Great Arteries (TGA) changes the incidence of major postoperative adverse events (AEs).

Major postoperative AEs include cardiac arrest, emergency chest opening, use of ECMO (machine that acts as an artificial heart and lung during surgery), and death.

Participants will be randomised to receive oxygen plus nitric oxide (intervention arm) or oxygen without nitric oxide (control arm) during CPB.

DETAILED DESCRIPTION:
The incidence of congenital heart disease (CHD) is approximately 1/100 live born children, of which up to 50% require cardiac surgery to correct the underlying abnormality at some stage during their life. (Centre for Disease Control and Prevention, USA). Despite major improvements in CPB devices, the exposure of host blood to large artificial organ surfaces, combined with myocardial injury during planned myocardial ischemia, results in a significant systemic inflammatory response. CPB-triggered systemic inflammatory syndrome is responsible for the most serious and potentially life-threatening side effects associated with cardiac surgery. It is characterized by endotoxin release, leukocyte and complement activation, and widespread activation of inflammatory mediators, resulting in endothelial leak, increased oxygen consumption, and organ dysfunction.

NO is an endogenous anti-inflammatory mediator that helps to protect endothelial beds and immunologically active cells. NO has a myocardial protective effect by reducing reperfusion injury. NO generation is essential for regulation of endothelial function and microvascular inflammation. However, dysregulation of endogenous NO during CPB may aggravate the subsequent inflammatory response.

A randomized controlled study adding NO into the bypass circuit was conducted by the Royal Children's Hospital in Melbourne on 198 children. This pilot study confirmed the positive effects of gaseous NO reported in the U.S. trial, as well as a reduction in the incidence of low cardiac output syndrome (LCOS). Other improved patient outcomes included a reduced need for extracorporeal life support (ECLS), trends towards a reduced length of stay, and shorter duration of ventilation. In light of these promising preliminary results from these two separate studies, a large multicentre trial to test these findings in children requiring cardiac surgery is needed.

The NASO study is running concurrently with the Nitric Oxide during Cardio Pulmonary Bypass during surgery for congenital heart defects: A Randomised Controlled Trial study (ANZCTR Trial Registry ID: ACTRN12617000821392) within Australia (run by Lady Cilento, Brisbane). This study is aiming to look at the effects of Nitric Oxide on all children under the age of 2 years undergoing bypass surgery for CHD.

TGA presents in 5-7% of all patients with congenital heart disease and isolated TGA is managed in a similar manner all over the world. The surgical treatment for this is the ASO. Hence this single operation and diagnosis provides an appropriate setting to evaluate the efficacy of NO in the CPB circuit. By allowing each centre to have their own protocols of care (pre, intra and postoperatively) and only collecting 'routine clinical data", the investigators anticipate each centre having high rates of screening and consent.

Patients will be stratified by centre and by age at time of surgery. Participants will be randomized into one of two arms:

* Intervention arm will receive NO 20 parts per million (ppm) into the oxygenator of a cardio-pulmonary bypass circuit
* Control arm will not receive NO

At the end of CPB, the participants will return to the Intensive Care Unit where normal care will continue.

A total of 800 participants will be enrolled in the study and will be stratified by centre and age at time of surgery.

Study aims to investigate whether exposure to gaseous NO reduces the incidence of postoperative major adverse events in infants on cardiopulmonary bypass.

ELIGIBILITY:
Inclusion criteria;

Each participant must meet all of the following criteria to be enrolled in this study:

* Infant aged greater than or equal to 36 weeks gestation
* Infants less than 2 years
* Diagnosed with TGA and requiring Arterial Switch Operation
* Consent of parents/guardian.

Exclusion criteria

Potential participants will be excluded if they meet any of the following criteria:

* They have multiple major congenital anomalies (anomalies which affect the infant's life expectancy or health status)
* They have multiple other cardiac abnormalities (with the exception of ASD, VSD or PDA)
* They weigh less than 2.2kgs.
* Prior surgical exposure to cardio-pulmonary bypass

Min Age: 0 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2018-07-11 (Actual); Primary Completion 2022-03-23 (Actual); Study Completion 2023-04-23 (Actual)

PRIMARY OUTCOMES:
Major adverse events | 28 days post intervention
  The primary outcome is the number of participants with major adverse events (MAEs) within 28 days post-operatively. MAEs include cardiac arrest, emergency chest opening, use of ECMO, and death.

SECONDARY OUTCOMES:
Length of stay in ICU (hours) | This will be calculated from date and time of admission to ICU to date and time of discharge from ICU in hours up to 28 days
  Length of stay in ICU (hours) will be calculated from date and time of admission to ICU date and time of discharge to ICU.
Length of stay in hospital (days) | 28 days (or until hospital discharge)
  Length of stay in hospital (days) will be calculated from date and time of admission to hospital to date and time of discharge to hospital.
Ventilator-free days | 28 days (or until ICU discharge)
  Ventilator-free days will be calculated from date and time of intubation to date and time of extubation. Each day (or part of a day) will be counted as a day.
Inotrope hours | Number of hours inotropes have been administered during first 28 days post operatively
  Inotrope hours will be calculated from data input into REDCAP.
Dialysis-free days | 28 days (or until ICU discharge)
  Dialysis-free days will be calculated from date and time of start of dialysis to date and time of stopping dialysis. Each day (or part of a day) will be counted as a day.
Inhaled NO hours | Number of hours inhaled NO have been administered during first 28 days post operatively
  Inhaled NO hours will be calculated from data input into REDCAP.
ECMO-free days | 28 days (or until ICU discharge)
  ECMO-free days will be calculated from date and time of start of ECMO to date and time of stopping ECMO. Each day (or part of a day) will be counted as a day.
Closed sternum days | 28 days (or until ICU discharge)
  Closed sternum days will be calculated from date and time of start of chest opening (or return to ICU time if delayed chest closure) to date and time of chest closure. Each day (or part of a day) will be counted as a day.
Composite free-day score | 28 days (or until hospital discharge)
  This score is a combination of scores 1-8 to create a composite free-day score. Composite free-day score is a score highlighting the number of days free from post-operative complications including free of hospitalization within the first 28 days post operatively. For each score, the days free of complication will be calculated to create an individual free from score these will be then added together to create an overall free-from score. Higher scores suggest a better outcome (free from hospital and complications).

CONTACTS AND LOCATIONS:
Overall Officials: Warwick Butt, Principal Investigator — MRCI
Locations (4):
- Royal Children's Hospital, Melbourne, Victoria, Australia
- Stollery Cildren's Hospital, Edmonton, Alberta, Canada
- Harapan Kita Children and Women's Hospital, Jakarta, Indonesia
- Institut Jantung Negara, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chello M, Mastroroberto P, Perticone F, Celi V, Colonna A. Nitric oxide modulation of neutrophil-endothelium interaction: difference between arterial and venous coronary bypass grafts. J Am Coll Cardiol. 1998 Mar 15;31(4):823-6. doi: 10.1016/s0735-1097(97)00560-3. PMID 9525554
- [Background] Hataishi R, Rodrigues AC, Neilan TG, Morgan JG, Buys E, Shiva S, Tambouret R, Jassal DS, Raher MJ, Furutani E, Ichinose F, Gladwin MT, Rosenzweig A, Zapol WM, Picard MH, Bloch KD, Scherrer-Crosbie M. Inhaled nitric oxide decreases infarction size and improves left ventricular function in a murine model of myocardial ischemia-reperfusion injury. Am J Physiol Heart Circ Physiol. 2006 Jul;291(1):H379-84. doi: 10.1152/ajpheart.01172.2005. Epub 2006 Jan 27. PMID 16443673
- [Background] Levy JH, Tanaka KA. Inflammatory response to cardiopulmonary bypass. Ann Thorac Surg. 2003 Feb;75(2):S715-20. doi: 10.1016/s0003-4975(02)04701-x. PMID 12607717
- [Background] Zahler S, Massoudy P, Hartl H, Hahnel C, Meisner H, Becker BF. Acute cardiac inflammatory responses to postischemic reperfusion during cardiopulmonary bypass. Cardiovasc Res. 1999 Mar;41(3):722-30. doi: 10.1016/s0008-6363(98)00229-6. PMID 10435044
- [Result] Checchia PA, Bronicki RA, Muenzer JT, Dixon D, Raithel S, Gandhi SK, Huddleston CB. Nitric oxide delivery during cardiopulmonary bypass reduces postoperative morbidity in children--a randomized trial. J Thorac Cardiovasc Surg. 2013 Sep;146(3):530-6. doi: 10.1016/j.jtcvs.2012.09.100. Epub 2012 Dec 8. PMID 23228403
- [Result] James C, Millar J, Horton S, Brizard C, Molesworth C, Butt W. Nitric oxide administration during paediatric cardiopulmonary bypass: a randomised controlled trial. Intensive Care Med. 2016 Nov;42(11):1744-1752. doi: 10.1007/s00134-016-4420-6. Epub 2016 Sep 30. PMID 27686343

DOCUMENTS (2):
  • Study Protocol (2019-01-25): https://cdn.clinicaltrials.gov/large-docs/85/NCT03661385/Prot_002.pdf
  • Informed Consent Form (2018-08-14): https://cdn.clinicaltrials.gov/large-docs/85/NCT03661385/ICF_001.pdf